CLINICAL TRIAL: NCT01393301
Title: Integrated Treatment for Smoking Cessation & Anxiety in People With HIV
Acronym: Project Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Southern Methodist University (Other); University of Houston (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Ph.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA031038-01A1 (NIH); 1R34DA031038-01A1 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nicotine Dependence; Symptoms of Anxiety; HIV
Keywords: Nicotine dependence; Smoking, cessation; Quitting; Anxiety symptoms; Cognitive-behavioral therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For formative stage of the study, no masking was used as that phase was an open pilot. Outcomes assessor masked during the pilot RCT.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Intervention Arm (Experimental): Standard smoking cessation treatment and nicotine replacement therapy (NRT) plus a cognitive-behavioral therapy for anxiety, depression, or other symptoms of distress.
  Interventions: Behavioral: Integrated cognitive-behavioral therapy for smoking cessation and anxiety
- Control Arm (Other): Enhanced Treatment as Usual (ETAU); enhanced standard smoking cessation treatment and nicotine replacement therapy (NRT).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Integrated cognitive-behavioral therapy for smoking cessation and anxiety — Standard smoking cessation treatment and nicotine replacement therapy (NRT) plus a cognitive-behavioral therapy for anxiety, depression, or other symptoms of distress.
  Other Names: QUESTT
  Arms: Behavioral Intervention Arm
Behavioral: Control — Enhanced standard smoking cessation treatment and NRT.
  Other Names: Enhanced Treatment as Usual (ETAU)
  Arms: Control Arm

SUMMARY:
During the 1-year formative phase of a study to develop an integrated treatment for quitting smoking for anxiety-vulnerable HIV+ smokers. During this first phase of the study, start-up activities will include piloting the integrated treatment on a small group of individuals (N = up to 12), obtaining expert consultant and participant feedback, and development of the final treatment manual and procedures. The goal during this phase will be to establish feasibility of treatment delivery, participant acceptability, and potential for a treatment effect before conducting a pilot randomized trial of the treatment. During the two-year pilot RCT phase of the above study, we directly develop and test a novel psychosocial/behavioral and pharmacological smoking cessation intervention for HIV+ smokers with interfering psychological distress.

DETAILED DESCRIPTION:
This study represents an important step in treating nicotine dependence in HIV-positive individuals. This study addresses an important public health issue by assessing an intervention that may lead to a more effective application for the treatment of at-risk HIV+ smokers. The 1-year formative phase of the study will develop an integrated treatment for quitting smoking for anxiety-vulnerable HIV+ smokers. The proposed treatment will include cognitive-behavioral talk therapy for quitting smoking, a nicotine patch, and cognitive-behavioral talk therapy for anxiety. The pilot of the proposed treatment will be conducted with a small group of individuals (N = up to 12). This phase will be used to establish feasibility of treatment delivery, and participant acceptability before conducting a pilot randomized trial of the treatment. Additionally, this phase will monitor smoking cessation history through Point Prevalence Abstinence (PPA), as well as anxiety symptoms through the Anxiety Sensitivity Index (ASI) at the baseline and follow-up assessments. This study represents an important step in treating nicotine dependence in HIV-positive individuals. This study addresses an important public health issue by assessing an intervention that may lead to a more effective application for the treatment of at-risk HIV+ smokers. The pilot RCT phase of the study (years 2 and 3), will test the developed cognitive-behavioral intervention in a pilot randomized-controlled trial format. The outcomes for this trial will be to determine the acceptability and feasibility of the intervention and the potential for an effect on increasing point prevalence abstinence and deceasing psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Informed consent
* Daily smoker
* Motivated to quit smoking

Exclusion Criteria:

* Use of other tobacco products
* Untreated or unstable psychiatric disorders
* Current use of cognitive-behavioral therapy or medication for smoking cessation treatment
* Insufficient command of English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conall O'Cleirigh, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] O'Cleirigh C, Zvolensky MJ, Smits JAJ, Labbe AK, Coleman JN, Wilner JG, Stanton AM, Gonzalez A, Garey L, Regenauer KS, Rosenfield D. Integrated Treatment for Smoking Cessation, Anxiety, and Depressed Mood in People Living With HIV: A Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2018 Oct 1;79(2):261-268. doi: 10.1097/QAI.0000000000001787. PMID 30212438

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 72 participants were officially consented, 71 participants completed baseline (1 lost to follow-up), and 53 participants attended Session 1 after baseline (10 found ineligible at baseline, 8 lost to follow-up). Randomization occurred at the end of Session 1; therefore, only participants who attended Session 1 (N=53) were randomized.
Period: Overall Study
Arm/Group | Behavioral Intervention Arm | Control Arm
Started | 26 | 27
Completed | 17 | 24
Not Completed | 9 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Completed <7 sessions (intervention) | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.73 (7.96) | 51.22 (8.54) | 50.49 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Treatment Acceptability
Description: Acceptability is defined as intervention participant study completion. Study completion was defined by participants attending at least 7/10 treatment sessions.
  Qualitative interviews were also conducted with participants at the end of the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Intervention Arm
Number analyzed (Participants) | 26
Participants | 17

2. Primary Outcome: Long-term Point Prevalence Abstinence (PPA; Pilot RCT Phase)
Description: Smoking outcomes are assessed at 6-month follow up by comparing the reported 7 day abstinence (assessed through self-report and independent verification) across the randomized conditions controlling for pre-randomization levels.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Intervention Arm | Control Arm
Number analyzed (Participants) | 13 | 21
Participants | 6 | 1

3. Primary Outcome: Short-term Point Prevalence Abstinence (PPA; Pilot RCT Phase)
Description: Smoking outcomes are assessed at end of treatment by comparing the reported 7 day abstinence (assessed through self-report and independent verification) across the randomized conditions controlling for pre-randomization levels.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Intervention Arm | Control Arm
Number analyzed (Participants) | 17 | 23
Participants | 10 | 2

4. Secondary Outcome: Treatment Related Changes in Psychological Distress.
Description: Treatment related changes in psychological distress was measured by combining the SIGH-A, MADRS, STAI-S, and CES-D into one scale score between baseline and the 6-month follow-up. In accordance with published recommendations, each psychological measure was z-scored to put all outcomes on the same scale. A z-score below 0 indicates a level of psychological distress below the mean (lower psychological distress), while a z-score above 0 indicates a level of psychological distress above the mean (higher psychological distress).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Behavioral Intervention Arm | Control Arm
Number analyzed (Participants) | 13 | 21
z-score | -.06 (.61) | .31 (.55)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Information was collected and reported for both study-related and non-study related adverse events.
Arm/Group | Behavioral Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/26 | 4/27
Other Adverse Events (participants affected / at risk) | 0/26 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention Arm (N=26) | Control Arm (N=27)
Hospitalization for dizziness (Endocrine disorders) | 1 (1) | 0 (0) — Participant hospitalized for feeling dizzy. After being released from hospital, participant engaged with their primary care provider and an endocrinologist.
Hospitalization for leg blockage (Cardiac disorders) | 0 (0) | 1 (1) — Participant experienced a leg blockage for which they were admitted to hospital for treatment.
Hospitalization for psychiatric reasons (Psychiatric disorders) | 0 (0) | 1 (1) — Participant experienced acute psychiatric symptoms and was hospitalized for treatment.
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalization for overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Accidental double dose of medication not related to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention Arm (N=26) | Control Arm (N=27)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Patient went to the emergency department for symptoms of pneumonia, but was not admitted to the hospital.
Intense Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Patient went to the emergency department due to symptoms of intense anxiety. Was not hospitalized, but the psychiatrist in the ED increased their anti-anxiety medication dosage.
Nicotine Patch Negative Effects (General disorders) | 0 (0) | 1 (1) — Within an hour of two of putting on nicotine patch for first time, patient experienced heart racing, vomiting, nausea, inability to leave bed, and thoughts/feelings of dread. Took off patch and symptoms subsided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No